CLINICAL TRIAL: NCT04104633
Title: Feasibility Study of a Molecular Karyotype Using a Very High-throughput Sequencing Approach, the "Massive Parallel Sequencing" on Circulating Tumor DNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Duffaut - Avignon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DEGENCA
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Colo-rectal Cancer
Keywords: ctDNA; Molecular karyotype
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with breast or colorectal cancer (Other): 10 patients with invasive breast carcinoma, not otherwise specified (NOS) (Stade I to III) and 10 patients with invasive colorectal adenocarcinoma (Stade I to III)
  Interventions: Procedure: Blood samples

INTERVENTIONS:
Procedure: Blood samples — 30 ml of blood collection

SUMMARY:
There are several types of circulating DNA: DNA from patient's existing cells, foetal DNA in the case of pregnant woman, and tumoral DNA in the case of patients with cancer. These circulating tumoral DNA (ctDNA) can be obtained from a blood test called liquid biopsy and be detected by the latest generation of very high throughput sequencers with the Massive Parallel Sequencing technique (MPS).

This study focus on using this technique on breast and colorectal cancers in which no analysis of CNV (tumor origin marker) with this technique has been performed yet. It is a prospective, pilot, monocentric, feasibility study on genomic profile. The study aim is to show the possibility to realize in a reproductive way a molecular karyotype on ctDNA with the MPS approach from a liquid biopsy taken from patients with cancer and to compare this profile with the one obtained by CGH array (Comparative Genomic Hybridization) from primitive tumor.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Signed consent
* Women with invasive breast carcinoma, NOS, with a radiologically measurable tumor of more than 10 mm (stade I to III)
* Patients with invasive colorectal adenocarcinoma with a radiologically measurable tumor of more than 10 mm (stade I to III)
* Patients who primary surgery is planned

Exclusion Criteria:

* Neoadjuvant chemotherapy or neoadjuvant radiotherapy
* Other cancer
* BMI > 30
* Pregnant woman
* Patients under protective administration or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of molecular karyotype performed from liquid biopsy: copies number variations (CNV) | Up to surgery
  Feasibility of molecular karyotype showing acquired copies number variations (CNV) on whole genome performed from ctDNA isolated from blood sample in patients with breast or colorectal cancer

SECONDARY OUTCOMES:
Identification of patient's tumor genomic profile with blood sample | Up to surgery
  Identification of patient's tumor genomic profile by comparison between genomic profile of primitive tumor obtained by CGH array and genomic profile of ctDNA obtained by Massive Parallel Sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume GRANIER, MD, Study Chair — Centre Hospitalier Henri Duffaut
Locations (1):
- Centre Hospitalier Henri Duffaut, Avignon, France

IPD SHARING:
Plan to Share IPD: No